CLINICAL TRIAL: NCT03731689
Title: Treatment of Intrauterine Adhesions and Its Distribution of Genital Tract Flora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuqing Chen, chief physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intrauterine adhesions
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Intrauterine Adhesions
Keywords: intrauterine lavage therapy; hysteroscopy; microbiome; uterine endometrial repair; intrauterine gel-injection therapy
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Control group( Intrauterine patients) do not apply intrauterine lavage therapy or intrauterine gel-injection therapy after surgery.
- Intrauterine lavage therapy group (Experimental): Intrauterine lavage therapy group apply intrauterine lavage therapy after surgery.
  Interventions: Drug: Intrauterine lavage therapy
- Intrauterine gel-injection therapy group (Experimental): Intrauterine gel-injection therapy group apply intrauterine gel-injection therapy after surgery.
  Interventions: Drug: Intrauterine gel-injection therapy
- Healthy control group (No Intervention): Healthy control group 1)have regular menstrual cycles,diagnostic hysteroscopy with endometrial biopsy and laparoscopy as part of their infertility diagnostic work-up prior to IVF, hysteroscopy and subsequent pathological results having shown no abnormality in the uterine cavities and abdominal cavity.2) had male partners who were infertile and diagnosed with defective sperm function,such as asthenozoospermia, oligoasthenozoospermia, severe oligoasthenozoospermia and azoospermia, defined according to guidelines published by the World Health Organization.

INTERVENTIONS:
Drug: Intrauterine lavage therapy — Intrauterine lavage treatment was performed within 3 to 7 days after the first menstrual period after surgery.
  Arms: Intrauterine lavage therapy group
Drug: Intrauterine gel-injection therapy — Intrauterine gel-injection treatment was performed within 3 to 7 days after the first menstrual period after surgery.
  Arms: Intrauterine gel-injection therapy group

SUMMARY:
This study aims to investigate the treatment of intrauterine adhesion and the factors influencing its prognosis.

DETAILED DESCRIPTION:
Intrauterine adhesion, also known as Asherman's syndrome, is the partial or complete occlusion of the uterine cavity as a result of endometrium damage. Most intrauterine adhesions patients manifest amenorrhea, reduced menstrual pattern, infertility, and intrauterine growth restriction, which seriously affect their reproductive health.It is well established that the formation of intrauterine adhesion likely involves hypoxia, reduced neovascularization, and altered expression of adhesion associated cytokines, but the exact mechanisms are not well understood. Although excessive curettage is considered the primary cause, intrauterine adhesion is known to be associated with diverse non-traumatic factors, such as postabortal sepsis, puerperal sepsis and infections. Intrauterine adhesion separation surgery is the gold standard for the treatment of uterine adhesion. Although the success rate is as high as 95%, the patients with moderate or severe uterine adhesion have severe damage to the endometrial basement, poor regeneration of endometrial and gland, poor tolerance of endometrial and poor clinical prognosis. Even if all kinds of anti-adhesion measures are used comprehensively, the postoperative recurrence rate of patients with moderate and severe uterine adhesion is high.Therefore this study was conducted to investigate whether intrauterine lavage or intrauterine gel-injection therapy after surgery could reduce the recurrence of intrauterine adhesion, promote the endometrial growth and repair and improve the menstruation and reproductive prognosis for severe intrauterine adhesion, and we hypothesize that intrauterine adhesion may be related to changes in microbial flora in the reproductive tract.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria(experimental group and control group):

* Pre-operative adhesion score was ≥5
* The prior menstrual cycle was regular, and the sex hormone was normal
* Patients had fertility requirement
* Male semen examination showed normal
* There were no severe systemic diseases, and no contradictions to aspirin, estrogen and surgery

Inclusion Criteria(healthy control group):

* regular menstrual cycles,diagnostic hysteroscopy with endometrial biopsy and laparoscopy as part of their infertility diagnostic work-up prior to IVF, hysteroscopy and subsequent pathological results having shown no abnormality in the uterine cavities and abdominal cavity
* the healthy women recruited had male partners who were infertile and diagnosed with defective sperm function,such as asthenozoospermia, oligoasthenozoospermia, severe oligoasthenozoospermia and azoospermia, defined according to guidelines published by the World Health Organization.

Exclusion Criteria:

* Pre-operative adhesion score was <5
* Prior menstrual cycle was irregular and sex hormone was abnormal, or patients had endocrine factors that caused amenorrhea, menstrual reduction and infertility
* Patients had no fertility requirement
* Patients(experimental group and control group) had male factor infertility
* Patients had contradictions to estrogen and aspirin such as cancers (breast cancer and endometrial cancer), thrombotic diseases, allergy to antipyretic analgesics, severe liver injury, hypoprothrombinemia, vitamin K deficiency, hemophilia, thrombocytopenia, gastric or duodenal ulcer and asthma.
* refuse Endometrial biopsy
* Vaginal discharge abnormal, or suspected vaginitis or pelvic inflammatory disease, or using antibiotics.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial Thickness of All Participants in the Mid Menstrual Measured by Color Doppler Ultrasound | 1 year

SECONDARY OUTCOMES:
Menstruation Pattern(Improvement or No Significant Change) of All Participants | 1 year
  A method similar to visual analogue scale(VAS) was employed for the evaluation of post-operative menstruation with 0 as amenorrhea and 100 as normal menstruation.
Reduction of American Fertility Society adhesion score at Second-look | one year
  The severity and extent of intrauterine adhesions were scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version) [7]. A score of 1-4 was considered to represent mild adhesions, a score of 5-8 was considered to represent moderate adhesions and a score of 9-12 represented severe adhesions.
Number of Participants With Pregnancy after operation | two years
Differences in distribution of reproductive tract bacteria between patients are before and after operation | one year
Differences in distribution of reproductive tract bacteria between healthy control group and intrauterine adhesion patients | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Chen, Deputy chief, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Guangzhou, Guangdong, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes